CLINICAL TRIAL: NCT02078336
Title: Optimization of Procedural Sedation Protocol Used for Dental Care Delivery in People With Mental Disability
Acronym: OptiSeDent
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: S55859; 2013-003991-11 (EudraCT Number)
Record Dates: First submitted 2014-02-24; First posted 2014-03-05 (Estimated); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Dental Care for Disabled
MeSH Terms: interventions — Diazepam; Biperiden; Droperidol; Atropine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Midazolam (Experimental): Midazolam Mylan 5 mg/ml solution for injection 15mg Oral use Single dose 45 minutes before dental treatment
  Interventions: Drug: Midazolam Mylan
- Lorazepam / Valium+Akineton+Dehydrobenzperidol+Atropine sulfat (Active Comparator): Lorazepam Mylan 2,5 mg tabletten 2.5mg Oral use Single dose 45 minutes before dental treatment
  OR
  Valium 10 mg/2 ml solution for injection 10mg Intramuscular use Single dose 45 minutes before dental treatment
  + Akineton 5 mg/ml solution for injection 5mg Intramuscular use Single dose 45 minutes before dental treatment
  + Dehydrobenzperidol 5 mg/2 ml solution for injection 0,000125 ml/cm2 Intramuscular use Single dose 45 minutes before dental treatment
  + Atropine sulfate Sterop 0,25mg/1ml solution for injection 0,25mg Intramuscular use Single dose 45 minutes before dental treatment
  Interventions: Drug: Lorazepam Mylan; Drug: Valium + Akineton + Dehydrobenzperidol + Atropine sulfate

INTERVENTIONS:
Drug: Midazolam Mylan
  Arms: Midazolam
Drug: Lorazepam Mylan
  Arms: Lorazepam / Valium+Akineton+Dehydrobenzperidol+Atropine sulfat
Drug: Valium + Akineton + Dehydrobenzperidol + Atropine sulfate
  Arms: Lorazepam / Valium+Akineton+Dehydrobenzperidol+Atropine sulfat

SUMMARY:
The study aims to compare procedural sedation protocols, specifically applied for the delivery of regular dental care in persons with a mental disability.

The primary objectives are:

* To assess the level of cooperation during regular dental care using different procedural sedation protocols
* To assess patient safety during regular dental care using different sedation protocols
* To assess patient comfort and possible side-effects after regular dental care using different sedation protocols

ELIGIBILITY:
Inclusion Criteria:

* Minimum age 18yrs
* Patient resides at least 6 months in nursing home "het Gielsbos".
* Patient always gets a sedative protocol to make dental care delivery possible.
* Informed consent was obtained from parent/guardian
* No medical contra-indication for any of tested sedative protocols

Exclusion Criteria:

* Age under 18yrs
* The patient is no resident of the nursing home "het Gielsbos" or lives there for less than 6 months.
* No need for medicinal support during dental treatment
* No informed consent was obtained by parents or the guardian of the patient.
* Medical contra-indication for 1 of the sedative protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-12; Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Level of cooperation of patient when receiving regular dental care | Participants will be followed for the duration of the dental treatment, an expected average of 30 minutes.

SECONDARY OUTCOMES:
Recording of vital parameters during regular dental care delivery | 24 hrs
  The measure is a composite of
  * recording of blood pressure
  * recording of pulse
  * recording of oxygen saturation
Level of patient comfort and possible side-effects after dental treatment session | 24 hrs
  The measure of patient comfort and possible side-effects after dental treatment session is a composite of
  * changes in appetite
  * changes in toilet behavior
  * changes in level of consciousness
  * changes in level of concentration
  * changes in pattern of epileptic insults
  * changes in mood
  * changes in sleeping pattern
  * changes in level of motor skills

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Declerck, Principal Investigator — KU Leuven
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Belgium